CLINICAL TRIAL: NCT04596956
Title: A Multicenter Randomized Controlled Trial on the Safety and Efficacy of Sodium Bicarbonate Ringer Injection in Elderly Patients Undergoing Abdominal Surgery
Brief Title: Safety and Efficacy of Sodium Bicarbonate Ringer Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director of the Center for Anesthesia, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020MZ01
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Ringer Bicarbonate; Elderly Abdominal Surgery; Safety; Effectiveness
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium bicarbonate Ringer injection (Experimental)
  Interventions: Drug: sodium bicarbonate Ringer injection
- Ringer lactate solution (Active Comparator)
  Interventions: Drug: Lactated Ringer's solution

INTERVENTIONS:
Drug: sodium bicarbonate Ringer injection — Used in surgery
  Arms: sodium bicarbonate Ringer injection
Drug: Lactated Ringer's solution — Used in surgery
  Arms: Ringer lactate solution

SUMMARY:
Objectives

1. To observe whether sodium bicarbonate Ringer injections can reduce the incidence of postoperative complications in elderly patients undergoing abdominal surgery.
2. To observe the effects of sodium bicarbonate Ringer injections on the internal environment, such as water, electrolytes, acid-base balance, and other physiological indexes, in the perioperative period of elderly patients undergoing abdominal surgery.

Research design：This study adopts a multicenter, prospective, randomized, controlled, pragmatic clinical trials (PCT) research design.

Sample size：5000 cases. Indication：The experimental group is the elderly patients undergoing abdominal surgery who were administered sodium bicarbonate Ringer injections intraoperatively; the control group is the elderly patients with abdominal surgery who were administered lactated Ringer's injections intraoperatively.

Observational index

Preoperative baseline data collection:

General patient information: basic information (age, height, and weight), preoperative diagnosis, past history, auxiliary examination results, etc.

Intraoperative data collection:

Perioperative vital signs information and arterial blood gas analysis results; The surgical method, operation time, and anaesthesia time; Intraoperative fluid management: The total amount of intraoperative fluids, blood transfusion volume, bleeding volume, urine volume, types and dosage of vasoactive drugs, diuretic dosage, sodium bicarbonate dosage.

Postoperative index:

Postoperative blood biochemical examination: liver function, renal function (urea nitrogen, creatinine), osmotic pressure, lactic acid, and blood sugar levels; Postoperative complications and treatment status Postoperative recovery: postoperative outcome, length of hospital stay, admission to ICU (duration of stay), postoperative eating time, out of bed activity time, gastrointestinal recovery time (exhaust), time for removal of various tubes (gastric tube, urinary tube, and drainage tube), etc.

The observation cut-off point is the patient's discharge. If the patient is still hospitalized 30 days after the operation, the observation will be terminated.

Research process

1. Elderly abdominal surgery patients who meet the inclusion criteria will be enrolled and randomly divided into two groups according to the intraoperative application of extracellular fluid supplements. The experimental group is sodium bicarbonate Ringer injection group, and the control group is sodium lactate Ringer injection. Basic preoperative information of patients will be collected. The vital signs, fluid treatment, and surgical anaesthesia will be recorded during the operation, while the recovery and postoperative complications will be recorded during postoperative visits.
2. The ability of sodium bicarbonate Ringer injections to reduce postoperative complications in elderly patients undergoing abdominal surgery will be observed.
3. The effects of sodium bicarbonate Ringer injection on the internal environment, such as water, electrolytes, acid-base balance, and other physiological indexes in elderly patients undergoing abdominal surgery will be observed and compared.
4. The safety and efficacy of sodium bicarbonate Ringer injection in elderly patients with abdominal diseases will be comprehensively assessed.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients need to be over 65 years of age, while there is no restriction on gender.
* (2) Patients are planned to undergo upper abdominal surgery under general anaesthesia, with an expected operation time of >2 h, and the infusion volume is >1000ml.
* (3) The patient agrees to participate in the clinical research and signs the informed consent.

Exclusion Criteria:

* (1) Emergency surgery
* (2) Hypermagnesemia (defined as serum Mg2+ >1.25mmol/L)
* (3) Patients who participated in other drug trials in the past 6 months
* (4) Known allergic reactions to the test drug and/or its components
* (5) Patients judged to lack the ability of providing informed consent
* (6) Other situations considered unsuitable for enrollment by the researcher.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Complication rate (including death) | 30days
  Complications include: bleeding, infection (incision infection, blood infection, urinary system infection), gastrointestinal complications (postoperative intestinal obstruction, anastomotic leakage), pulmonary complications (pulmonary infection, pulmonary embolism) ), cardiovascular complications (cardiac arrest, arrhythmia, heart failure, myocardial infarction), neurological complications (delirium, stroke), urinary system complications (renal insufficiency), etc. (refer to International Surgical Prognosis Study, ISOS ), and died during hospitalization.

IPD SHARING:
Plan to Share IPD: Undecided